CLINICAL TRIAL: NCT01917942
Title: A Randomised Phase III Trial of Radiotherapy With Humidification in Head And Neck Cancer
Brief Title: Radiotherapy With Humidification in Head And Neck Cancer
Acronym: RadioHum
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Collaborators: Auckland City Hospital (Other Government); Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TROG 07.03; NCT00598520 (obsolete NCT alias)
Record Dates: First submitted 2013-08-01; First posted 2013-08-07 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Cancer of the Head and Neck
Keywords: Radiotherapy; Humidification; Mucositis
MeSH Terms: conditions — Head and Neck Neoplasms; Mucositis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care (Active Comparator): Standard of Care
  Interventions: Other: Standard of Care
- Humidification (Experimental): Humidification
  Interventions: Device: Humidification

INTERVENTIONS:
Device: Humidification — Fisher and Paykel Healthcare MR880 humidifier + HC211 flow source. 37/44 Humidification (37oC at 100% relative humidity, 44 mg of water per litre of air, 25 litres per min initial flow rate). The patients will be instructed to use humidification from day 1 of the radiotherapy course as much as is practical; the preference is for continuous overnight humidification plus maximal use throughout the day.Humidification will continue throughout treatment until at least week 8 after the commencement of radiotherapy and will cease when the CTCAE mucositis (clinical exam) score becomes less than grade 2, or at the week 16 assessment, whichever is earliest.
  Arms: Humidification
Other: Standard of Care — SOC: institutional standard of care for the management of mucositis. SOC will be defined by each participating institution and be kept consistent at that institution for the duration of the study. In general, SOC will consist of rinsing with 50:50 salt bicarbonate of soda mouthwash; benzydamine mouthwash; appropriate analgesic, antimicrobial and antifungal protocols etc.
  Arms: Standard of Care

SUMMARY:
This is a two arm randomised phase III trial which will evaluate prospectively the benefits of humidification in patients receiving radiotherapy / chemoradiation for head and neck cancer. The intent of humidification is to moisturise the mucosa. The rationale for the use of humidification with radiotherapy can be considered an extension of the general principle of moist wound care in wound management.

DETAILED DESCRIPTION:
This phase III trial will address four hypotheses. The primary hypothesis is:

Humidification will modulate the natural history of mucositis resulting in a clinically significant reduction in the intensity of severe acute mucositis as a function of time for CTCAE grade > 1 mucositis (e.g. grade 2 or higher), measured as the area under the time curve (AUC) of the plot expressing grade of acute reactions vs weeks for observed CTCAE mucosal reactions > 1

The additional hypotheses are:

* Humidification will palliate the acute symptoms of mucositis and xerostomia
* Humidification is cost effective through a reduction in hospital bed occupancy
* Humidification will improve the functional outcome, particularly swallowing function, of patients with head and neck cancer treated with radiotherapy

ELIGIBILITY:
Inclusion Criteria:

Patients who meet the following criteria will be eligible:

* Pathologically confirmed diagnosis of cancer involving the Nasopharynx, Oropharynx, Oral Cavity, Larynx, or Hypopharynx
* Regional nodal irradiation included in PTV1 (as a minimum ipsilateral levels II-III)
* Prescribed dose of radiotherapy is at least 60 Gy
* Receiving definitive or post-operative adjuvant Radiotherapy
* Receiving Radiotherapy as sole modality or Chemoradiation
* Patient > 18 years old
* Available for follow-up for up to 2 years
* Life expectancy greater than 6 months
* Written informed consent
* Participation of patients on other clinical trial protocols permitted

Exclusion Criteria:

Patients who meet the following criteria will be excluded:

* Presence of tracheostomy or stoma
* Diagnosis of T1 / T2 glottic carcinoma
* Undergoing CPAP therapy -Treatment with Amifostine or Palifermin (keratinocyte growth factor) during radiotherapy
* History of previous radiotherapy to the head and neck region, excluding superficial radiotherapy to cutaneous squamous cell carcinoma or basal cell carcinoma
* High risk for poor compliance with radiotherapy, humidification, or follow-up as assessed by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2008-06; Primary Completion 2011-11 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Intensity of mucositis as a function of time for CTCAE grade > 1 mucositis (e.g. grade 2 or higher) measured as the area under the time curve (AUC) of the plot expressing grade of acute reactions vs weeks for observed CTCAE mucosal reactions > 1. | week 12

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Macann, Study Chair — Auckland Hospital
Locations (1):
- Auckland Hospital, Auckland, New Zealand

REFERENCES:
- See also: Click here for more information about this study on the TROG official website — http://www.trog.com.au